CLINICAL TRIAL: NCT03942861
Title: Sonographic Assessment in Severe Ulcerative Colitis Patients Admitted for Intravenous Corticosteroids and Eligible for Infliximab Rescue Therapy; a Prospective Clinician-blinded Observational Study Protocol.
Acronym: SUCCES
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Copenhagen University Hospital at Herlev (Other)
Responsible Party: Principal Investigator, Johan F. Ilvemark, MD, Principal Investigator, Copenhagen University Hospital at Herlev
Other Study IDs: CopenhagenUHH
Record Dates: First submitted 2019-04-25; First posted 2019-05-08 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Ulcerative Colitis; Ultrasound Therapy; Complications
Keywords: Ultrasonography; Sonography; Ulcerative Colitis; Inflammatory Bowel Disease; Severe Ulcerative colitis; Treatment response; Monitoring treatment
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — Methylprednisolone Hemisuccinate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Severe Ulcerative Colitis: Consecutive patients admitted as in-patients to the Department of Gastroenterology at four University Hospitals in Denmark, with acute severe UC defined as an affirmed diagnosis of UC according to well established criteria, combined with a Mayo score of 8 or more (i.e. severe disease activity) and the need for intravenous corticosteroid treatment will be screened for participation in the study after informed consent.
  Interventions: Drug: Solu-Medrol

INTERVENTIONS:
Drug: Solu-Medrol — Standard treatment according to Danish Guidelines for acute severe ulcerative colitis.

SUMMARY:
Introduction Acute severe ulcerative colitis (ASUC) occurs in 15-25 % of all ulcerative colitis (UC) patients. Initial treatment with intravenous corticosteroids fails in 30-50 % of patients, for whom the next line of treatment is biological therapy or colectomy. Acute colectomy has a higher risk of morbidity and mortality than a scheduled colectomy. Data suggest that an accelerated administration of biological treatment in corticosteroid non-responders compared to clinical practice, 5-7 days with intravenous corticosteroids, may be superior in inducing disease remission, thus potentially avoiding acute colectomy. However, there are currently no patient friendly and objective diagnostic tool to preselect patients for such a treatment. The aim of this study is to examine if gastrointestinal ultrasound (GIUS) could preselect corticosteroid non-responders to biological treatment after 48 hours to increase effectiveness of the second line therapy and thereby reduce the morbidity and mortality of ASUC.

Methods and analysis The study is a clinician blinded observational multi-center study derived from the Department of Gastroenterology, Herlev Hospital, Denmark. Fifty ASUC patients will be included at the time of hospitalization and followed for 12 months. Baseline clinical activity scores, endoscopic scores, blood samples, fecal-calprotectin, vital parameters and GIUS measurements will be obtained prior to administration of intravenous corticosteroids. All examinations except fecal-calprotectin and endoscopy will be repeated at 48 ± 24 hours, 5-7 days and 3 months after treatment start. Endoscopic scores and fecal-calprotectin will be obtained after 3 months and an additional fecal-calprotectin after 6 ± 1 days. Treatment outcome will be registered at each event and after 12 months. Patients will be divided into corticosteroid responders and non-responders and compared to GIUS measurements at each event using non-parametric statistics (Mann-Whitney and Wilcoxon test) and time to endpoints by survival statistics (Kaplan Meier). ROC statistics will determine the best cutoff values for GIUS parameters for optimal sensitivity, specificity and accuracy.

Ethics and dissemination The study is approved by the National committee on health research ethics (H-18031264). Results will be published in relevant scientific journals and presented at international conferences. Fully anonymized data will be accessible from authors upon request.

DETAILED DESCRIPTION:
Introduction

Ulcerative colitis (UC) is a chronic inflammatory bowel disease (IBD), typically diagnosed between the age of 15 and 40 and characterized by colonic mucosal inflammation and ulcerations. These mucosal changes lead to bloody diarrhea and in severe cases, fever, anemia, weight loss and death if not treated appropriately. The condition requires prompt immunosuppressive treatment and monitoring. To characterize disease severity and guide treatment decisions, clinicians typically use a combination of clinical scores based on patients symptoms, endoscopic scoring systems based on mucosal appearance endoscopic assessments of disease extent and blood and stool markers of inflammation.

Most patients experience a mild to moderate disease course with varying periods of activity and remission. However, 15-25 % will experience a flare of acute severe UC (ASUC), a condition characterized by extensive and deep ulcerations on endoscopy combined with a high clinical score of severity. Due to the risk of bowel wall perforation, these patients are usually admitted to the hospital ward for intensive monitoring and medical therapy. The medical therapy ultimately aims at avoiding acute colectomy, a procedure that still carries a 30-day mortality rate of 5 %, which is higher compared to elective surgery (OR 1.82; CI 95 % 1.19 - 2.62). Initial therapy is well established and consists of intravenous corticosteroids, which in early clinical trials dramatically improved the disease outcome by reducing the mortality rate from 24 to 7 %. Unfortunately, even today 30 - 50 % of patients with ASUC fails to respond to initial corticosteroid treatment and are therefore eligible for medical rescue treatment if surgery is not imminent.

Accordingly, primary non-responders to high dose intravenous corticosteroids are usually switched to infliximab (or at certain centers ciclosporine) after 5-7 days, if an acute colectomy is not needed. Infliximab is an anti-tumor necrosis factor (TNF) alpha antibody, which blocks TNFα, a key inflammatory mediator in UC,and has been proven effective in corticosteroid resistant UC reducing the risk of acute colectomy from 58 % to 29 %.

Despite advances in medical treatment ASUC still carries a 10 % risk of acute colectomy. Further improvement in medical therapy and strategy is therefore highly warranted. A decrease in serum albumin is associated with an increased clearance of infliximab, and it has been suggested that postponement of infliximab treatment in ASUC could reduce the bioavailability of the drug as a result of severe hypoalbuminemia. In addition, infliximab is lost in feces in the setting of ASUC, suggesting that an accelerated infliximab induction regimen or an increased starting dose compared to standard procedures could be beneficial. However, a recent review of retrospective studies showed no difference in colectomy rates when comparing an accelerated infliximab induction regimen with standard induction regimen (both induced after 3-5 days of corticosteroid treatment), although confounding by disease severity cannot be excluded. Hence it is currently unresolved if optimized timing and dosing of infliximab rescue treatment could be of major importance to reduce the need of acute colectomies and thereby the morbidity and mortality among ASUC patients. Therefore, data to support clinician's recognition of corticosteroid non-responders early in the process are warranted.

Unfortunately, there are currently no patient friendly, effective or objective point-of-care tool to identify corticosteroid non-responders early in the process. A high clinical score, C-reactive protein (CRP) and a low albumin is correlated with an inferior response, but due to poor positive and negative predictive values they are not routinely used to pre-select patients for specific medical therapies. Endoscopic severity is predictive for the outcome of ASUC, but the use of close monitoring with endoscopy is limited in this setting due to the risk of perforation and the need for repeated bowel cleansing.

Transabdominal gastrointestinal ultrasound (GIUS) is potentially a relevant objective point-of-care tool, which could be used for treatment outcome assessment in ASUC. A recent study in ulcerative colitis patients using GIUS to monitor anti-TNFα treatment demonstrated a high correlation between change in GIUS parameters, bowel wall thickness (BWT) and color Doppler Signal (DS), compared to baseline with treatment response after 6 and 12 weeks. The results are in accordance with other studies showing a correlation between endoscopic activity, clinical symptom scores, CRP and GIUS parameters after 2-3 months of treatment. In this setting, GIUS can also predict treatment outcome after 12-15 months. Ultrasound has several advantages compared to other modalities as it is non-invasive and does not inflict pain, is easily repeatable and available and does not expose the patient to radiation. Although some studies suggest 4 hours of fasting to diminish peristalsis and intraluminal air, fasting before examination is generally not necessary, making it preparation free.

Not all bowel segments can be easily visualized, which can be an issue when assessing disease extent. Especially the rectum and the left colonic flexure can be difficult to visualize and examine with the transabdominal approach. The combined reported sensitivity and specificity for detection of colonic inflammation is 74 % and 93 % per segment, whereas the sigmoid colon and the terminal ileum are easy to identify and measure, showing a higher diagnostic performance (sensitivity 92 % and specificity 87 %) compared to endoscopy. There is no significant difference in diagnostic accuracy per bowel segment compared to other radiologic modalities and in the latest ECCO guidelines GIUS is recommended as a valid alternative to CT or MR.

There are different signs of inflammation to look for when examining the bowel using GIUS; the most reported and prominent one being BWT. BWT in healthy subjects ranges between 0.5-3.0 mm depending on anatomical location. Studies on UC patients use different cutoff values, usually ranging between 3.0-4.0 mm. There is an ongoing discussion within the scientific community about cutoff values. In general, sensitivity decreases and specificity increases with a higher value. Vascularization is another important measure and can be estimated with DS and the Limberg score to define the presence of a high blood flow; a high blood flow correlates well with inflammation. Further, the bowel wall layers are easily identified due to echo-stratification on ultrasound. These layers are still present in the mild and moderate UC cases, whereas the stratification can be lost in severe UC. Severe inflammation can also cause colonic de-haustration, although this parameter might also correlate to the chronicity of the condition. Inflammatory mesenteric fat wrapped around the affected intestine is rarely seen in UC patients but frequently in Crohn's disease.

No study examining the ability of GIUS to predict treatment response in ASUC patients has yet been conducted on a shorter timeframe than 6 weeks. The investigators have unpublished preliminary data suggesting a rapid detectable change in GIUS parameters in patients responding to high-dose corticosteroids. If GIUS can be used as an objective point-of-care tool for treatment response, it may be useful to identify corticosteroid non-responders at an early stage, thus providing an opportunity for optimized individual treatment, i.e. rescue infliximab treatment, and hopefully a decreased morbidity and mortality rate.

Methods and analysis

Study aims The primary aim is to determine if early changes in GIUS parameters (BWT, vascularization, echostratification, inflammatory mesenteric fat and haustration) from baseline to 48 ± 24 hours after intravenous corticosteroids initiation in hospitalized patients with ASUC, can predict clinical corticosteroid non-response and need for biological treatment and/or colectomy.

The secondary aims are to:

1. Determine if changes in GIUS parameters from baseline to day 6 ± 1 and 3 months after intravenous corticosteroids initiation can predict treatment non-response and need for colectomy.
2. Identify the potential interrater variability between investigators and central reading for GIUS parameters.
3. Correlate GIUS parameters with changes in fecal calprotectin and endoscopic disease activity (Mayo endoscopic sub-score and Ulcerative Colitis Endoscopic Index of Severity (UCEIS)) at baseline and 3 months after hospitalization.
4. Correlate GIUS parameters with changes in clinical scores (Mayo score and Simple Clinical Colitis Activity Index (SCCAI)), blood samples (hemoglobin, CRP, albumin and alpha-1-antitrypsin), pulse, blood pressure, temperature and time since last meal at 48 ± 24 hours, 6 ± 1 days and 3 months after hospitalization.
5. Examine GIUS´s ability to assess disease extent compared to endoscopy and CT (if a CT-scan is performed after an ordination by a treating physician).
6. Determine the ideal cutoff values for GIUS parameters for optimal sensitivity, specificity and accuracy.

Study design The study design is a prospective clinician blinded multi-center observational study. Fifty patients will be included and followed for 12 months. The study is approved by the Danish National committee on health research ethics H-18031264 and the Danish data protection agency VD-2018-319.

Procedures and scheduled follow-up visits

Included patients will prior to intravenous corticosteroid treatment have the following information registered as baseline characteristics:

* Date of birth, age at disease diagnoses, previous and present IBD medication, previous intestinal surgery, previous extent of disease, other known chronic diseases, smoking status, extra-intestinal manifestations, weight and height, symptoms (blood and frequency of stools, urgency of defecation, general well-being, physician's general assessment), family history of IBD and previously known gastrointestinal infections (Clostridium difficile, Salmonella, Campylobacter jejuni, CMV, Yersinia enterocolitica or other).
* Mayo endoscopic sub-score, UCEIS and current endoscopic extent of inflammation.
* Blood samples (hemoglobin, CRP, albumin, alpha - 1 - antitrypsin), fecal calprotectin results, pulse, blood pressure and temperature.
* GIUS assessment of the BWT, vascularization, echostratification, inflammatory mesenteric fat and haustration.
* Time since last meal prior to GIUS examination. The intestinal ultrasound together with blood samples and recordings of pulse, blood pressure, temperature, time since last meal, time since first intravenous corticosteroid administration as well as clinical scores will be repeated 48 ± 24 hours, 6 ± 1 days and 3 months after the first dose of intravenous corticosteroids. Endoscopic examination and fecal calprotectin will be repeated after 3 months. Treatment outcome (response to corticosteroid, infliximab or colectomy) will be registered at 48 ± 24 hours, 6 ± 1 days, 3 months and 12 months after the first dose of intravenous corticosteroids. Results of eventual CT-scans or extra endoscopies will be stored.

Clinical assessment Patient disease status is monitored during hospitalization using the Mayo clinical score and SCCAI. Mayo clinical score is based on blood and stool frequency, baseline endoscopy results and the physician's global assessment. SCCAI is based on bowel frequency divided by night and day, urgency of defecation, blood in stool, patient general well-being and extra-intestinal features. Endoscopic severity is graded using the Mayo endoscopic subscore and the UCEIS, which is based on the severity of the vascular pattern, presence of blood, erosions and ulcers. The clinical assessment and endoscopies will be performed by a physician blinded to the GIUS measurements. Endoscopic assessment is based on the worst segment and documented with still images on a secure drive.

GIUS assessment and measurements Each examination will be performed by a GIUS trained gastroenterologist using the same high-end ultrasound scanner and 9L probe for the same patient. Probe frequency will be between 5-8 MHz. Scans are performed by localizing the sigmoid colon at the site of the iliac vessels and then followed in both anal and oral direction. The most severe part of the bowel segment will be assessed and documented by still images and cineloop files and stored in DICOM format on a secure drive. Sigmoid colon is always assessed as the primary point of interest. However, if topical treatment has been applied or a more oral located bowel segment has a higher BWT this segment will also be documented as above and stored. GIUS examination recordings will be subjected to central reading by an independent GIUS specialist, blinded to the original scans. Fasting will not be required, but the time passed since patients last meal will be registered. The GIUS examiner will have no knowledge about the patient disease status (blood and stool sample results, clinical scores or endoscopic activity).

• BWT is measured in the most severe segment (largest BWT) using the average value of four measurements with one decimal (two longitudinal scans, more than 1 cm apart and two cross-sectional scans, which can be in the same image, but in different quadrants). A BWT value < 3.0 mm is regarded as no inflammation and ≥ 3.0 mm is regarded as active disease.

In segments with a BWT ≥ 3.0 mm, vascularization will be classified using a color Doppler and a modified Limberg score, as well as echostratification and the eventual presence of inflammatory mesenteric fat and absence of haustration.

* Vascularization is measured in both the cross-sectional and longitudinal plane. Pathological vascularization is defined as a modified Limberg score > 1 and normal vascularization is defined as ≤ 1. No signal, 0 points; minimal pixels, 1 point; increased doppler signal limited to the wall, 2 points; and if the signal is significant in the wall as well as the mesentery, 3 points.
* Normal echostratification is measured in a longitudinal plane and defined as 3-5 echo layers in each bowel wall (mucosa, submucosa, lamina muscularis) and will be characterized as 1. normal/preserved, 2. uncertain, 3. focal disruption < 3 cm or 4. extensive disruption ≥ 3 cm.
* Inflammatory mesenteric fat will be defined as a bright looking mass surrounding or wrapping the bowel, usually brighter and more homogenous than normal intraabdominal fat in obese; characterized as either 1. absent, 2. uncertain or 3. present.
* Haustration will be defined as either 1. present (normal), 2. uncertain or 3. absent.

Centre selection The study is devised by leading researchers in IBD and trained bowel ultrasound experts at the Department of Gastroenterology, Herlev Hospital, Denmark. The IBD clinic at Herlev Hospital is one of the largest clinical and academic IBD centers in Denmark and an international training center for GIUS. Recruitment and examination of the patients will be conducted at the gastroenterological departments of the university hospitals in Herlev, Aarhus, Vejle and Hvidovre. All GIUS gastroenterologists engaged in the study meet and train together to make the procedures identical and standardized before patient inclusion.

Sample size calculation The sample size was calculated to be able to detect a 0.7-fold decrease in thickness of the intestinal wall with a common standard deviation (sigma) of 30 % and a desired power of 80 % to determine a statistically significant difference (α = 0.05, two-sided test). The estimated sample size is 17 subjects in each group (responders/non-responders). The investigators aim to include 20 UC patients in each group, and since 40 % are expected to be non-responders to steroids, the overall aim is to include 50 patients. Our department currently admits 3-5 patients/month with ASUC. Together with the other departments, the estimated inclusion period is 15 months.

Statistical analysis Clinical data will be entered into a validated data capture system provided by the Danish Capital Region. The data system will include password protection and internal quality checks, such as automatic range checks, to identify data that appear inconsistent, incomplete or inaccurate. Descriptive data will be provided for all outcomes (table 2) according to data type; number of patients, mean, SD (for interval data), median 25 % and 75 % quartiles (for ordinal data). Frequency (absolute and relative) distributions will be provided for categorical data. Two-sided p values will be presented throughout. Data management and analysis will be performed using REDCap and SPSS.

Primary endpoint analysis Patients will be divided into steroid responders and steroid non-responders and compared to GIUS parameters (BWT, modified Limberg score, echostratification, inflammatory mesenteric fat and haustration at baseline to 48 ± 24 hours) using non-parametric statistics (Mann-Whitney and Wilcoxon test) and time to endpoints by survival statistics (Kaplan Meier).

Secondary endpoints analysis The same statistical tests as used for primary endpoint analysis will be applied to predict responders versus non-responders throughout the observational period. GIUS measurements at baseline compared to 6 ± 1 days and 3 months, with a follow up at 12 months. GIUS interrater-variability between GIUS examiners and proof reader will be calculated as kappa values, interclass correlation co-efficiency and Limits of Agreement for continues variables. Correlation between the GIUS measurements and endoscopic variables will be assessed using Spearman's rank correlation coefficient, multiple logistic regression and receiver operating characteristics (ROC) analyses. An additional ROC analyses will be performed to determine the best cutoff values for GIUS parameters for optimal sensitivity, specificity and accuracy.

Variables associated with non-responders and responders GIUS measurements (CRP, Hemoglobin, Albumin, alpha-1-antitrypsin, Mayo clinical score, SCCAI, pulse, blood pressure, temperature, time since last meal and fecal calprotectin) will be assessed with univariate analyses. Those who achieve a p-value of < 0.2 will be included into a multivariable logistic regression analysis.

Discussion There is an unfulfilled need for a reliable, easy, non-invasive and safe modality to repeatedly assess treatment response in patients admitted with ASUC. GIUS presents itself as such a modality and the investigators hypothesize that within 48 hours after corticosteroid treatment GIUS has the potential to identify steroid non-responders. This has not previously been investigated. An early identification allows for an accelerated treatment decision in steroid resistant ASUC patients and thus a potential decrease in the need of acute colectomies. To achieve this goal, the investigators first need to validate GIUS as a point-of-care tool to predict treatment outcome in patients with ASUC.

Ethics and dissemination In accordance with the Helsinki V declaration and the Ethics committee of the Capital Region of Denmark enrollment in the study is based on voluntary informed written consent. All patients can at any time withdraw their participation without any change in standard care or treatment. Written information about the project will ensure patient knowledge of their rights. Ultrasound is a safe and patient friendly examination without any side effects, damage or radiation for the patient. The trial will contribute to a new partially unexplored field with promises of improving disease activity monitoring and consequently more rational and timely treatment intervention and decreased morbidity and mortality. Results will be published in international journals and disseminated at international conferences.

ELIGIBILITY:
Inclusion Criteria:

* Definitive diagnoses of Ulcerative colitis.
* Mayo clinical score ≥8.
* Need for Hospitalization and intravenous corticosteroid treatment.
* Age between 18-70.
* Ability and willingness to give written consent and comply with study protocol.

Exclusion Criteria:

* Contraindicators for infliximab.
* Bowel infection.
* Crohn's disease.
* Ultrasonographic inflammation in terminal ileum other than backwash ileitis.
* Bowel wall thickness <3 in Sigmoid colon.
* Minors.
* Known malignant disease.
* Pregnancy.
* Immune modulating therapy at admission apart from corticosteroids, mesalazine or azathioprine.

Contraindicators = Patients suffering from moderate to severe heart failure, hypersensitivity to murine proteins, severe bacterial infection.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Consecutive patients admitted as in-patients to the Department of Gastroenterology at four University Hospitals in Denmark, with ASUC defined as an affirmed diagnosis of UC according to well established criteria, combined with a Mayo score of 8 or more (i.e. severe disease activity) and the need for intravenous corticosteroid treatment will be screened for participation in the study after informed consent.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-02-21 (Actual); Primary Completion 2021-09-21 (Estimated); Study Completion 2022-02-21 (Estimated)

PRIMARY OUTCOMES:
Changes in GIUS parameters 48 hours after intravenous corticosteroid treatment. | The outcome measure will be assessed after 18 months and reported within 36 months.
  Number of patients stratified by treatment response (defined by a decrease in clinical Mayo score from baseline ≥ 30 % and ≥ 3 points, along with either a rectal bleeding subscore of 0 or 1 or a decrease in rectal subscore ≥ 1 point) and non-response and their respective change in GIUS parameters (BWT, modified Limberg score, echostratification, inflammatory mesenteric fat and haustration) at 48 ± 24 hours after corticosteroid treatment compared to baseline.

SECONDARY OUTCOMES:
Changes in GIUS parameters ability to predict treatment outcome. | The outcome measure will be assessed after 18 months and reported within 36 months.
  Number of patients stratified after treatment response and non-response after 6 ± 1 days, within 3 months and after 12 months compared to changes in GIUS parameters at each event compared to baseline.
Interrater variability compared to central reading with regards to GIUS parameters. | The outcome measure will be assessed after 18 months and reported within 36 months.
  All GIUS scans will be performed by a trained GIUS gastroenterologist and proof read by a second specialist. We wish to examine eventual differences between their assessments.
Time since last meal correlated to feasibility of GIUS. | The outcome measure will be assessed after 18 months and reported within 36 months.
  Although some studies suggest 4 hours of fasting to diminish peristalsis and intraluminal air, fasting before examination is generally not necessary, making it preparation free. We will register patients time since last meal and correlate it to feasibility of GIUS.
GIUS disease extent assessment compared to endoscopy and CT (if present). | The outcome measure will be assessed after 18 months and reported within 36 months.
  Number of correct GIUS assessment of inflammatory extension compared to endoscopy and CT (if present), which is seen as the golden standard, defined by location (rectum, sigmoid colon, descending colon, transverse colon, ascending colon and terminale ileum.
Calculate the best cutoff value for GIUS parameters for optimal sensitivity, specificity and accuracy compared to treatment outcome and endoscopy results. | The outcome measure will be assessed after 18 months and reported within 36 months.
  ROC analyses will be performed to determine the best cutoff values for GIUS parameters for optimal sensitivity, specificity and accuracy in predicting treatment outcome (responder vs. non-responder).
Change in GIUS parameters correlation with change in endoscopic scores and fecal calprotectin within 3 months compared to baseline. | The outcome measure will be assessed after 18 months and reported within 36 months.
  Change in GIUS parameters for steroid responders and non-responders and correlation with change in Mayo endoscopic sub-score, UCEIS and fecal calprotectin within 3 months compared to baseline.
Change in GIUS parameters correlation with change clinical scores and biochemistry on 48 ± 24 hours, 6 ± 1 days and after 3 months compared to baseline. | The outcome measure will be assessed after 18 months and reported within 36 months.
  Change in GIUS parameters for steroid responders and non-responders and correlation with change in Mayo clinical score, SCCAI, CRP, alpha-1-antitrypsin and increase of albumin or hemoglobin on 48 ± 24 hours, 6 ± 1 days and after 3 months compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Jakob B. Seidelin, MD, PhD, Principal Investigator — Copenhagen University Hospital at Herlev
Locations (1):
- Herlev University Hospital, Copenhagen, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Our plan is that fully anonymized data will be accessible from authors upon request.